CLINICAL TRIAL: NCT00503919
Title: A Pilot Study: Measurement of Digital Colposcopy for Fluorescence Spectroscopy of the Normal Cervix for Screening, Using a Second Generation Device
Brief Title: Measurement of Digital Colposcopy for Fluorescence Spectroscopy of TNC Using a Second Device
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed early with no enrollment.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-0810
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2009-09

CONDITIONS: Cervical Neoplasia
Keywords: Cervix; Cervical dysplasia; Cervical neoplasia; Cervical intraepithelial neoplasia; Multi-spectral Digital Colposcopy; MDC; Acetic acid; Colposcopy; Spectroscopy; Fluorescence Spectroscopy; Abnormal Pap Smear
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDC (Experimental): Multi-spectral Digital Colposcopy for Fluorescence Spectroscopy
  Interventions: Procedure: Multi-spectral Digital Colposcopy (MDC)

INTERVENTIONS:
Procedure: Multi-spectral Digital Colposcopy (MDC) — Use of a digital camera and a special light to take pictures of the cervix and vagina.

SUMMARY:
The overall objective of this study is to identify potential improvements for a noninvasive method of diagnosing dysplasia and neoplasia in the cervix using Multi-spectral Digital Colposcopy (MDC), a device that uses fluorescence and reflectance spectroscopy to compare images to histopathologic mapping of the cervical epithelium.

Primary Objective:

-To measure Multi-spectral Digital Colposcopy images in vivo of the cervix both before and after acetic acid in a screening population.This is a second generation research device with low significant risk for which we are studying MDC.

Secondary Objectives:

1. To evaluate the effect of the fading of acetic acid in the image contrast obtained over time to see if this fading can predict the presence of any neoplasia.
2. To evaluate mapping the cervix so that software can reconstruct the cervical epithelial map as evaluated by a Papanicolaou Smear to compare to routine colposcopic images as well as those from the Multi-spectral Digital Colposcopy (MDC).

DETAILED DESCRIPTION:
A colposcopy is an exam of the vagina and cervix using a magnifying lens. A multi-spectral digital colposcopy uses a digital camera and a special light to take pictures of the cervix and vagina.

Before taking part in this study, you will have a complete medical history recorded. You will have a physical exam and a pap smear. Women who are able to have children must have a negative urine pregnancy test.

You will then have a multi-spectral digital colposcopy performed during the routine colposcopy in the outpatient clinic. A multi-spectral digital colposcopy device will shine light on the cervix and vagina and take several pictures. The pictures will be used by the doctors to check the cells and structure of the tissue. After the first set of pictures, acetic acid (vinegar) will be applied to the cervix so any lesions would show up better. Application of acetic acid is a normal part of the colposcopy and not part of the research. About 1-2 minutes later, more pictures will be taken.

If the acetic acid/colposcopy show abnormal cells, you will have a biopsy of the cervical canal.

If the acetic acid /colposcopy show normal cells, no biopsy will be taken.

Once you have completed the colposcopy with or without the biopsy of the cervical canal, your participation on this study is complete.

If either your Pap smear or biopsy of the cervical canal is abnormal, the study doctor/staff will recommend further care or treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years of age or older.
2. Women who have been referred for screening at U.T.M.D. Anderson Hospital, Houston, TX USA; U.T. Health Science Center-Houston,TX USA; Lyndon B. Johnson General Hospital, Houston, TX USA; British Columbia Cancer Agency, Vancouver, British Columbia, Canada; and the University College Hospital, Ibadan, Oyo State, Nigeria, Africa Cervical Screening Clinics, Family Planning Clinics or Gynecology Clinics.
3. Patients must sign an informed consent indicating awareness of the investigational nature of the study.

Exclusion Criteria:

1. Patients will be considered ineligible if they are pregnant.
2. If they have a history of an abnormal Pap or a treatment to the cervix.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal cell detection before and after acetic acid/colposcopy using Multi-spectral Digital Colposcopy (MDC) | Participation limited to Colposcopy visit, anticipate study completion in one day
  Measurements of normal sites during colposcopy before and after the application of acetic acid using Multi-spectral Digital Colposcopy (MDC) images in vivo of the cervix both before and after acetic acid. Three images (white, blue, and green light) compared before and after acetic acid placement, the images may be compared to pathology obtained from a Pap Smear taken to evaluate the performance of the instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Milbourne, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org